CLINICAL TRIAL: NCT00125047
Title: Effectiveness of a Combined Vi Vaccination and Health Education Program on Reducing the Burden of Typhoid During Childhood: A Demonstration Project in Karachi
Brief Title: Combined Vi Vaccination and Health Education Program on the Burden of Typhoid in Childhood
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Aga Khan University (Other); Wellcome Trust (Other); University of Western Ontario, Canada (Other); GlaxoSmithKline (Industry)
Responsible Party: Mr. Leon Ochiai, International Vaccine Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: T-7
Record Dates: First submitted 2005-07-28; First posted 2005-07-29 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Typhoid; Paratyphoid Fever
Keywords: Salmonellosis; typhoid vaccine; enteric fever
MeSH Terms: conditions — Typhoid Fever; Paratyphoid Fever; Salmonella Infections | interventions — Vi polysaccharide vaccine, typhoid; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Typhoid Vi polysaccharide vaccine
  Interventions: Biological: Typhoid Vi vaccine
- 2 (Active Comparator): Inactivated Hepatitis A vaccine
  Interventions: Biological: Hepatitis A vaccine

INTERVENTIONS:
Biological: Typhoid Vi vaccine — Single 0.5ml dose containing 25ug purified Vi polysaccharide of S. typhi.
  Other Names: Typherix
  Arms: 1
Biological: Hepatitis A vaccine — single 0.5ml dose contains 720 EL.U. of inactivated hepatitis A viral antigen
  Other Names: Havrix
  Arms: 2

SUMMARY:
This study is part of the International Vaccine Institute's (IVI's) typhoid Vi demonstration project that aims to accelerate the rational introduction of Vi vaccines in typhoid endemic countries. The purpose of this study is to determine the effectiveness of the Vi vaccine following a mass typhoid immunization campaign in an endemic area in Karachi, Pakistan. The cost-effectiveness of Vi vaccination and the logistic feasibility of a mass typhoid immunization campaign will also be evaluated.

DETAILED DESCRIPTION:
Typhoid fever is a major cause of morbidity worldwide. The disease predominantly affects school-aged children, is more prevalent in urban areas, may last for several weeks and can lead to serious complications. Management of this disease is further complicated by the emergence of multi-drug resistant strains. Vaccination of high risk populations is considered the most promising strategy for the control of typhoid fever. The Vi polysaccharide vaccine has been targeted for accelerated introduction into public health programs due to the following reasons: it has been shown to have consistent efficacy results even in areas of high typhoid incidence; is given as a single dose; lacks patent protection and requires less strict cold chain requirements. A cluster-randomized trial involving the Vi polysaccharide vaccine and an active control (hepatitis A) was designed to determine the effectiveness and the feasibility of providing Vi vaccine under actual programmatic conditions in 3 urban slums in Pakistan. The vaccines used in this study are internationally produced and locally licensed. A complimentary, targeted, basic typhoid prevention health education program for the entire population at the initiation of the project will be provided and the actual Vi-demonstration project will be preceded by a 12-month typhoid surveillance activity.

Secondary objectives of this trial are:

* To monitor the adverse events following a routine Vi mass vaccination campaign;
* To assess the knowledge, attitudes, beliefs and practices among parents and health care providers regarding typhoid illness, treatment and prevention; and
* To study typhoid fever risk factors in the population.

A nested, prospective matched case-control study is included in the trial in order to study typhoid risk factors among children in Karachi.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the project census
* Age: 2-16 years

Exclusion Criteria:

* Fever >37.5 degrees Celsius, axillary
* Pregnancy
* Lactating

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27231 (Actual)
Dates: Start 2001-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Total protection against S. typhi | 2 years from zero time

SECONDARY OUTCOMES:
Indirect protection against s. typhi | two years from zero time
Overall protection against s. typhi | 2 years from zero time
Adverse event(s) following immunization | 30 days from vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, MBBS, PhD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Pakistan

REFERENCES:
- [Background] Ali M, Rasool S, Park JK, Saeed S, Ochiai RL, Nizami Q, Acosta CJ, Bhutta Z. Use of satellite imagery in constructing a household GIS database for health studies in Karachi, Pakistan. Int J Health Geogr. 2004 Sep 28;3(1):20. doi: 10.1186/1476-072X-3-20. PMID 15450121
- [Background] Acosta CJ, Galindo CM, Ochiai RL, Danovaro-Holliday MC, Page AL, Thiem VD, Park JK, Park E, Koo H, Wang XY, Abu-Elyazeed R, Ali M, Albert MJ, Ivanoff B, Pang T, Xu ZY, Clemens JD. The role of epidemiology in the introduction of vi polysaccharide typhoid fever vaccines in Asia. J Health Popul Nutr. 2004 Sep;22(3):240-5. PMID 15609776